CLINICAL TRIAL: NCT05535270
Title: Psychometric Properties of the Oxford Depression Questionnaire in Chinese Patients With Mood Disorders
Brief Title: Validation of the Chinese Version of Oxford Depression Questionnaire
Status: Completed | Type: Observational
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Principal Investigator, Hu ShaoHua, Head of Department of Psychiatry, First Affiliated Hospital of Zhejiang University, First Affiliated Hospital of Zhejiang University
Other Study IDs: IIT20220240B-R1
Record Dates: First submitted 2022-09-06; First posted 2022-09-10 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2023-09

CONDITIONS: Mood Disorders; Emotional Blunting
MeSH Terms: conditions — Mood Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Mood Disorder patients: The participants completed a demographic questionnaire, the self-report Oxford Depression Questionnaire (ODQ-C), the Beck Depression Inventory-II(BDI-II), and the Montgomery-Asberg Depression Rating Scale (MADRS).
  Interventions: Diagnostic Test: Oxford Depression Questionnaire (ODQ)
- Healthy Controls: The participants completed a demographic questionnaire, Patient Health Questionnaire - 9(PHQ-9), and the first two sections of Oxford Depression Questionnaire (ODQ-20).
  Interventions: Diagnostic Test: Oxford Depression Questionnaire (ODQ)

INTERVENTIONS:
Diagnostic Test: Oxford Depression Questionnaire (ODQ) — The Oxford Depression Questionnaire (ODQ)is a patient-centered questionnaire. The scale contains three sections: i) the patient's experience in the past week; ii) the patient's experience before the illness worsened, and iii) the patient's emotional feelings about receiving antidepressant treatment. The 26-item questionnaire contains four dimensions of "emotional blunting": not caring (NC), emotional detachment from others (ED), reduction in positive emotions (RP), and general reduction in emotions (GR). Patients not taking antidepressants were only required to rate the first two sections .

SUMMARY:
Mood disorders are a group of psychiatric disorders that can affect a person's mood, energy, and motivation. Emotional blunting has been observed in clinical practice in patients with mood disorders. Emotional blunting has a negative impact on patients' overall treatment and leads to poorer adherence. The Oxford Depression Questionnaire (ODQ) is a measuring instrument of emotional blunting. The ODQ is expected to be a scientifically valid tool for detecting emotional blunting. The ODQ has high construct validity and internal reliability. However, no scientific validity studies have been conducted on ODQ in Chinese population. Therefore, this study is intended to investigate the reliability and validity of the ODQ in Chinese patients with mood disorders.

ELIGIBILITY:
Inclusion Criteria:

1) both biological parents were Han Chinese; 2) currently diagnosed with major depressive disorder or bipolar disorder according to the Mini International Neuropsychiatric Interview for Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition; 3) aged 13-65 years; 4) can complete the self-assessment questionnaires.

Exclusion Criteria:

1) currently diagnosed with neurological diseases or other major psychiatric disorders, e.g., schizophrenia, cognitive impairment, substance abuse; 2) diagnosed with severe somatic illnesses, such as diabetes and cardiovascular diseases;

Ages: 13 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Participants with mood disorders are recruited as outpatients or inpatients with the First Affiliated Hospital of Zhejiang University, School of Medicine.
Sampling Method: Non-Probability Sample
Enrollment: 272 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Oxford Depression Questionnaire (ODQ) | baseline
  To analyze reliability and validity of the ODQ.

SECONDARY OUTCOMES:
Beck Depression Inventory-II (BDI-II) | baseline
  To analyze criterion validity of the Chinese version of the ODQ
Montgomery-Asberg Depression Rating Scale (MADRS) | baseline
  To analyze correlation with ODQ
Oxford Depression Questionnaire (ODQ) | 2 weeks after baseline
  To analyze Test-retest reliability coefficients of the ODQ.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Psychiatry, First Affiliated Hospital of Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No
Arms and interventions can be shared, while the clinical data will not be shared